CLINICAL TRIAL: NCT05988801
Title: Clinical and Radiographic Evaluation of Glass Ionomer Sealant Versus Resin Sealant for Pits and Fissures of the First Permanent Molars: A Randomized Clinical Trial.
Brief Title: Evaluation of Glass Ionomer Sealant Versus Resin Sealant for Pits and Fissures of the First Permanent Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abrar Hossam Ahmed Saleh, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Glass Ionomer VS Resin sealant
Record Dates: First submitted 2023-07-13; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pits and Fissures Sealant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glass ionomer sealant (Experimental): glass ionomer based sealant material
  Interventions: Other: Glass ionomer sealant
- Resin sealant (Active Comparator): resin-based sealant material
  Interventions: Other: Resin based sealant

INTERVENTIONS:
Other: Glass ionomer sealant — glass ionomer-based sealant material
  Arms: Glass ionomer sealant
Other: Resin based sealant — resin-based sealant material
  Arms: Resin sealant

SUMMARY:
evaluation of the clinical and radiographic success of the glass ionomer sealant versus resin sealant in the pits and fissures sealing of the first permanent molars

DETAILED DESCRIPTION:
GIC has a hydrophilic nature which makes it compatible with clinical situations when isolation may be difficult. It also sets rapidly, which can reduce sensitivity to moisture. Glass ionomers release fluoride, which promotes enamel remineralization and has an antimicrobial effect. Another benefit of using glass ionomers as sealants is that the tooth does not need to be etched to achieve chemical bonding to the tooth. Thus saving time which is critical in the case of young patients and patients with disabilities.

ELIGIBILITY:
Inclusion Criteria:

* • Children aged between 6 to 9 years

  * Children with deeply stained fissures of the first permanent molars.
  * First permanent molars are completely erupted
  * The patient's willingness to receive treatment

Exclusion Criteria:

* • Special child, a child with compromised systemic health.

  * First permanent molars covered by operculum.
  * Children with high salivary flow when isolation will be impossible

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Marginal discoloration | 6 months
  Marginal discoloration will be measured with visual examination and recorded in Alfa: Lack of discoloration, Bravo: Margin discoloration, and Charlie: Discoloration under the sealant.

SECONDARY OUTCOMES:
sealant retention | 6 months
  Sealant retention will be measured with a mouth mirror and probe and recorded in total retention or partial loss or complete loss
Dental Caries | 6 months
  The absence or presence of any signs of dental caries or periapical infection will be measured with a periapical X-ray

IPD SHARING:
Plan to Share IPD: No